CLINICAL TRIAL: NCT05779371
Title: Effects of the Integrated-based Laughing Qigong Program on Resilience in Community-dwelling Older Adults: An Explanatory Sequential Mixed Method
Brief Title: Effects of the Integrated-based Laughing Qigong Program on Resilience in Community-dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, Ph.D., RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: FJU-IRB C106177
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Community-dwelling Older Adults
Keywords: resilience, Integrated-based Laughing Qigong Program

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded to group membership, research assistants collected data from both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Experiment group A accepted the Integrated-based Laughing Qigong Program (IB-LQP) During the intervention, the participants formed a standing circle and could make eye contact. The time was divided into 10 minutes of warm-up (deep breathing, stretching of muscles, expressing various emotions on the face, stretching of limbs) and 30-40 minutes of main exercise (Breathing and Laughing Qigong practice). The main exercise included using the natural breath of laughter to activate the body, turning a fake smile into a real smile and laughter, using different body movements at the same time, producing a variety of types of laughter, and conducting self-emotional awareness and emotional transformation drills to reduce the backlog.
  Interventions: Behavioral: Integrated-based Laughing Qigong Program
- control group (No Intervention): The control group received no intervention and was asked to maintain their current lifestyle for 6 weeks following the baseline test.

INTERVENTIONS:
Behavioral: Integrated-based Laughing Qigong Program — The protocol of the Integrated-based Laughing Qigong Program (IB-LQP) combined laughter intervention and mental health promotion courses. It was a two-hour community activity held twice a week for six weeks. The content was 50-60 minutes of a laughter practice program and 50 minutes of mental health lectures, separated by a 10-minute break.
  Arms: Experimental group

SUMMARY:
Laughter programs are safe, affordable, and age-appropriate activities. Few studies have utilized mixed study designs to look at the impact on resilience in and experiences of participants in such activities.

DETAILED DESCRIPTION:
A high level of resilience can also help to mitigate the negative effects of stress and promote personal adaptation. According to a prior study, the resilience scale can be used to screen and identify maladaptive people before they cause problems, allowing for the development of preventive interventions (Wells, 2012). Some researchers have used cross talk and laughter therapy in patients with depression and reported that the negative symptoms of their mental health were alleviated (Yoshikawa et al., 2019), and laughter therapy for disabled adolescents improved their resilience (Shinde, & Kotekar, 2022). Another researcher discovered through interviews that older adults who laugh can maintain their personal health and age successfully (Lewis, 2021), but there is currently little research on how laughter affects the resilience of older adults.

Previous research applied laughter as a mental health-promoting activity, called the Laughter Qigong program, to promote mental health and generate positive effects on both physical and mental well-being (Hsieh et al., 2015). According to Kuru Alc, Zorba Bahceli, and Emirolu (2018), laughter intervention is risk-free, inexpensive, and beneficial for promoting the mental health of older adults. It has been used successfully with these people in long-term care facilities (Hsieh et al, 2015). The IB-LQP was administered twice weekly for four weeks to older adults living in institutions. It was discovered to have a positive impact on stress cortisol levels (Hsieh et al., 2015), as well as the ability to lessen death fear and enhance loneliness (Kuru Alc, Zorba Bahceli, & Emirolu, 2018). The research on laughter-based interventions for community senior citizens is still in its early stages, and more research is needed to fully understand how senior citizens participate in locally tailored activities.

ELIGIBILITY:
Inclusion Criteria:

(1) age of ≧ 65 years, (2) ability to travel to the location of the activities on their own (independent or partially dependent people with daily activities), and (3) willingness to participate in this activity intervention

Exclusion Criteria:

(1) Severe hearing or sensory deficits that cause communication barriers, (2) diagnosis of depression, and (3) hospitalization plans in the next three months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 39 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Chinese Version of the Resilience Scale | Pre-intervention(T0)
  The content of the Chinese version of the Resilience Scale includes five levels: a meaningful life, a peaceful mind, self-confidence, an indomitable spirit, and acceptance of the loneliness of existence. The highest score is 7 points (extremely satisfied), and the lowest score is 1 point (extremely dissatisfied). A higher score indicates greater resilience (Ahern, Kiehl, Sole, and Byers, 2006). Psychometric assessment of this scale has supported its internal consistency reliability and concurrent validity as good, and many studies have confirmed that the scale is applicable to samples of all ages and races (Ahern, Kiehl, Sole, Byers, 2006). The Cronbach's α for internal consistency in this study was .91.
The Face Scale | Pre-intervention(T0)
  The face scale is a nonverbal emotion scale used to evaluate students' participation in courses (Lorish and Maisiak, 1986). It has seven faces, with number one representing the happiest and number seven representing the saddest. Before and after taking the " IB-LQP " course, the participants chose the facial scale that best represented their mood. This scale is appropriate for assessing emotions after older adults participate in activities and has high reliability (Hsieh et al., 2015).
Chinese Version of the Resilience Scale | 6-week after intervention (T1)
  The content of the Chinese version of the Resilience Scale includes five levels: a meaningful life, a peaceful mind, self-confidence, an indomitable spirit, and acceptance of the loneliness of existence. The highest score is 7 points (extremely satisfied), and the lowest score is 1 point (extremely dissatisfied). A higher score indicates greater resilience (Ahern, Kiehl, Sole, and Byers, 2006). Psychometric assessment of this scale has supported its internal consistency reliability and concurrent validity as good, and many studies have confirmed that the scale is applicable to samples of all ages and races (Ahern, Kiehl, Sole, Byers, 2006). The Cronbach's α for internal consistency in this study was .91
The Face Scale | 6-week after intervention (T1)
  The face scale is a nonverbal emotion scale used to evaluate students' participation in courses (Lorish and Maisiak, 1986). It has seven faces, with number one representing the happiest and number seven representing the saddest. Before and after taking the " IB-LQP " course, the participants chose the facial scale that best represented their mood. This scale is appropriate for assessing emotions after older adults participate in activities and has high reliability (Hsieh et al., 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Chia Jung Hsieh, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bath PA, Deeg D. Social engagement and health outcomes among older people: introduction to a special section. Eur J Ageing. 2005 Mar;2(1):24-30. doi: 10.1007/s10433-005-0019-4. Epub 2005 Mar 9. No abstract available. PMID 28794713
- [Result] Ahern NR, Kiehl EM, Sole ML, Byers J. A review of instruments measuring resilience. Issues Compr Pediatr Nurs. 2006 Apr-Jun;29(2):103-25. doi: 10.1080/01460860600677643. PMID 16772239
- [Result] Bahari, K., & Lorica, J. D. 2019. The effects of laughter therapy on mental health: An integrative literature review. The Malaysian Journal of Nursing (MJN), 10(3), 55-61. https://doi.org/10.31674/mjn.2019.v10i03.008
- [Result] Crane MF, Searle BJ, Kangas M, Nwiran Y. How resilience is strengthened by exposure to stressors: the systematic self-reflection model of resilience strengthening. Anxiety Stress Coping. 2019 Jan;32(1):1-17. doi: 10.1080/10615806.2018.1506640. Epub 2018 Aug 1. PMID 30067067
- [Result] Dyer JG, McGuinness TM. Resilience: analysis of the concept. Arch Psychiatr Nurs. 1996 Oct;10(5):276-82. doi: 10.1016/s0883-9417(96)80036-7. PMID 8897710
- [Result] Ellis JM, Ben-Moshe R, Teshuva K. Laughter yoga activities for older people living in residential aged care homes: A feasibility study. Australas J Ageing. 2017 Sep;36(3):E28-E31. doi: 10.1111/ajag.12447. Epub 2017 Jul 12. PMID 28699684
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] Fetters MD, Curry LA, Creswell JW. Achieving integration in mixed methods designs-principles and practices. Health Serv Res. 2013 Dec;48(6 Pt 2):2134-56. doi: 10.1111/1475-6773.12117. Epub 2013 Oct 23. PMID 24279835
- [Result] Fontes AP, Neri AL. Resilience in aging: literature review. Cien Saude Colet. 2015 May;20(5):1475-95. doi: 10.1590/1413-81232015205.00502014. English, Portuguese. PMID 26017950
- [Result] Hsieh CJ, Chang C, Tsai G, Wu HF. Empirical study of the influence of a Laughing Qigong Program on long-term care residents. Geriatr Gerontol Int. 2015 Feb;15(2):165-73. doi: 10.1111/ggi.12244. Epub 2014 Feb 18. PMID 24533887
- [Result] Ketefian S. Ethical considerations in research. Focus on vulnerable groups. Invest Educ Enferm. 2015;33(1):164-72. doi: 10.17533/udea.iee.v33n1a19. PMID 26148168
- [Result] Kilpatrick LA, Siddarth P, Milillo MM, Krause-Sorio B, Ercoli L, Narr KL, Lavretsky H. Impact of Tai Chi as an adjunct treatment on brain connectivity in geriatric depression. J Affect Disord. 2022 Oct 15;315:1-6. doi: 10.1016/j.jad.2022.07.049. Epub 2022 Jul 26. PMID 35905792
- [Result] Kuru Alici N, Zorba Bahceli P, Emiroglu ON. The preliminary effects of laughter therapy on loneliness and death anxiety among older adults living in nursing homes: A nonrandomised pilot study. Int J Older People Nurs. 2018 Dec;13(4):e12206. doi: 10.1111/opn.12206. Epub 2018 Jul 13. PMID 30004172
- [Result] Kirmayer LJ, Pedersen D. Toward a new architecture for global mental health. Transcult Psychiatry. 2014 Dec;51(6):759-76. doi: 10.1177/1363461514557202. Epub 2014 Oct 30. PMID 25358524
- [Result] Kuiper, N.A. (2012). Theoretical Contributions Humor and Resiliency: Towards a Process Model of Coping and Growth. Europe's Journal of Psychology, 2012, Vol. 8(3), 475-491, doi:10.5964/ejop. v8i3.464
- [Result] Lewis, J. P. 2021. The role of laughter in the resilience and wellbeing of Alaska native elders. In The Routledge International Handbook of Indigenous Resilience (pp. 208-221). Routledge. DOI: 10.4324/9781003048428-18
- [Result] Li SYH, Bressington D. The effects of mindfulness-based stress reduction on depression, anxiety, and stress in older adults: A systematic review and meta-analysis. Int J Ment Health Nurs. 2019 Jun;28(3):635-656. doi: 10.1111/inm.12568. Epub 2019 Jan 17. PMID 30656813
- [Result] Lorish CD, Maisiak R. The Face Scale: a brief, nonverbal method for assessing patient mood. Arthritis Rheum. 1986 Jul;29(7):906-9. doi: 10.1002/art.1780290714. PMID 3741503
- [Result] Madsen W, Ambrens M, Ohl M. Enhancing Resilience in Community-Dwelling Older Adults: A Rapid Review of the Evidence and Implications for Public Health Practitioners. Front Public Health. 2019 Feb 7;7:14. doi: 10.3389/fpubh.2019.00014. eCollection 2019. PMID 30792974
- [Result] Mertens, D.M. and Hesse-Biber, S. (2012). Triangulation and Mixed Methods Research: Provocative Positions. Editorial. Journal of Mixed Methods Research 6(2) 75-79 DOI: 10.1177/1558689812437100